CLINICAL TRIAL: NCT05439083
Title: Immunogenicity of 9-valent HPV Vaccine in Immunocompromised Children and Adolescents
Brief Title: Immunogenicity of 9-valent HPV Vaccine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Talia Sainz Costa (Other)
Responsible Party: Sponsor-Investigator, Talia Sainz Costa, Principal Investigator, Instituto de Investigación Hospital Universitario La Paz
Organization: Instituto de Investigación Hospital Universitario La Paz (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19042021/22
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Human Papilloma Virus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Two groups of patients:
  Immunosuppressed Group: N=90 Immunosuppressed patients, consisting of HIV-infected children and adolescents, hematopoietic stem cell transplant (HSCT) recipients, solid organ transplant (SOT) recipients and post-chemotherapy patients (PCT) under follow-up at Hospital La Paz in Madrid Spain.
  Control Group: N=30 Healthy controls aged 9-14. Both groups receive the 9-valent HPV vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunosuppressed Group (Experimental): N=90 Immunosuppressed patients, consisting of HIV-infected children and adolescents, hematopoietic stem cell transplant (HSCT) recipients, solid organ transplant (SOT) recipients and post-chemotherapy patients (PCT) under follow up at Hospital La Paz in Madrid Spain.
  9-valent HPV vaccine: three-dose schedule: Months 0-2-6.
  Interventions: Biological: 9-valent HPV vaccine
- Control Group (Other): N=30 Healthy controls aged 9-14 9-valent HPV vaccine: two-dose schedule: Months 0-6.
  Interventions: Biological: 9-valent HPV vaccine

INTERVENTIONS:
Biological: 9-valent HPV vaccine — All participants will receive the immunization schedule according to guidelines: immunosuppressed patients will receive a three-dose schedule: 0.5 mL intramuscular injection of 9vHPV at entry plus an additional dose at month 2 and month 6. Healthy controls aged 9-14 years will receive a two-dose schedule: 0 and 6 months.

SUMMARY:
Human papillomavirus (HPV) causes the most prevalent sexually transmitted infections in the world. The nonavalent HPV vaccine (9vHPV) provides protection against 9 high-risk HPV serotypes, responsible for causing approximately 90% of cervical and other HPV-related anogenital cancers, as well as 90% of genital warts. The risk of cancer is substantially increased among immunocompromised patients.

Although studies have demonstrated seroprotection among children and adolescents, boys and girls, with the 9vHPV vaccine, the immunogenicity of this vaccine has been poorly explored in immunocompromised children and adolescents (including transplant patients, and those infected with human immunodeficiency virus (HIV)). Several factors, including the immunological consequences of vertically acquired infection, immunosuppressive therapies and age, could lead to an increased risk of infection in children and adolescents who are immunocompromised. Lower immunogenicity in these populations. These children may have a poor response to vaccines and therefore require additional doses. Markers such as CD4/CD8 or torque teno virus (TTV) replication could be linked to immunogenicity and thus serve as predictors of efficacy for routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents 9 to <18 years of age
* Willing to sign consent/assent form
* If HIV positive, under ART and undetectable viral load and CD4 cell count >200/mm3 (at least 6 months)
* If the patient has received chemotherapy or is a SOT/HSCT recipient, referred for immunizations after adequate immune reconstitution according to routine clinical practice

Exclusion Criteria:

* Previous history of warts and/or anal cancer.
* Previous immunization with any HPV vaccine.
* Age below 9.
* Patients who for any reason should not be included in the study according to the evaluation of the research team.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Seroconversion of subjects from baseline to month 7 (determined by serum anti-HPV antibody titers) | From baseline to month 7
  Percentage of subjects seroconverting from baseline to month 7
Seroconversion of subjects from baseline to month 12 (determined by serum anti-HPV antibody titers) | From baseline to month 12
  Percentage of subjects maintaining antibody titers 12 months after immunization.
Seroconversion of subjects from baseline to month 18 (determined by serum anti-HPV antibody titers) | From baseline to month 18
  Percentage of subjects maintaining antibody titers 18 months after immunization.

SECONDARY OUTCOMES:
Ratio of geometric mean serum antibody titers (GMTs) | From baseline to month 7
  GMTs from baseline to month 7
Delta of geometric mean serum antibody titers | From 1 to 12 months
  Delta of geometric mean serum antibody titers from 1 to 12 months after immunization.
Percentage of subjects seroconverting from baseline to month 7 | From baseline to month 7
  Percentage of subjects seroconverting from baseline to month 7 in each of the study populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La paz, Madrid, Spain